CLINICAL TRIAL: NCT05867654
Title: Oral Versus Intravenous Antibiotics for the Management of the Osteomyelitis of the Jaws: An Open-Label Non-Inferiority Single-Arm Clinical Trial
Brief Title: Efficacy of Oral vs IV Antibiotics in the Treatment of Orofacial Osteomyelitis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: Osteo Science Foundation (Unknown)
Responsible Party: Principal Investigator, Suzanne Barnes, Assistant Professor, DMD, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22.0386
Record Dates: First submitted 2023-01-20; First posted 2023-05-22 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Osteomyelitis of Jaw
MeSH Terms: interventions — Amoxicillin-Potassium Clavulanate Combination; Clindamycin; Levofloxacin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Osteomyelitis Treated with Oral Antibiotics (Other): Patients that are receiving oral antibiotics for the treatment of their osteomyelitis.
  Based on the indication, patients will receive one the following medications orally for 6-8weeks: Amoxicillin-clavulanate 875mg/125mg q12hrs, clindamycin 300mg q6hrs, Levofloxacin 750mg QID, Penicillin 500mg q6hrs
  Interventions: Drug: Amoxicillin-clavulanate 875mg/125mg q12hrs; Drug: oral clindamycin 300mg q6hrs; Drug: Levofloxacin 750mg QID

INTERVENTIONS:
Drug: Amoxicillin-clavulanate 875mg/125mg q12hrs — Oral antibiotic used based on indication
  Other Names: Augmentin
Drug: oral clindamycin 300mg q6hrs — Oral antibiotic used based on indication
  Other Names: Cleocin
Drug: Levofloxacin 750mg QID — Oral antibiotic used based on indication
  Other Names: Levaquin

SUMMARY:
The goal of this clinical trial is compare the efficacy of oral and IV antibiotics in the treatment of orofacial osteomyelitis. The main question it aims to answer is: Are oral antibiotics as effective as IV antibiotics in the treatment of orofacial osteomyelitis.

Participants, once diagnosed with osteomyelitis, will be started on oral antibiotics for their treatment. Participants will follow up with oral and maxillofacial surgery clinic accordingly and their progression and compliance will be monitored.

DETAILED DESCRIPTION:
We plan to conduct a randomized controlled open label trial of PO versus IV antibiotics in treatment of patients with osteomyelitis of the jaws. The clinicians caring for the patient will decide what antibiotics to give to the patient and the route or antibiotic therapy will be oral unless this route of administration fails and the patient does not wish to extend the oral antibiotics route. After thorough discussion of the risks, benefits, and alternatives, a consent form is reviewed and signed. The clinicians' choice of antibiotic prescribed will be according to the common practices and standards, with modifications, when necessary, based on local antibiotic guidelines, and in consultation with Infectious Disease (ID) team at our institute when needed. Participants will include patients with osteomyelitis of the jaws diagnosed by the Oral and Maxillofacial Surgery (OMFS) Department of the University of Louisville for eligibility. We will determine if the patient meets the inclusion and exclusion criteria, and, if the patient is willing, a study member will obtain informed consent. If patients provide informed consent, we will then record the clinical diagnosis and demographic data. These forms will be stored in our clinic and scanned in patient's medical records for future reference. We will see the patients according to our routine schedule in our clinic. This schedule includes the primary consultation appointment, admission, and inpatient surgery, the first follow-up 24-72 hours after discharge from hospital, one week follow up afterwards, and then follow-ups at two weeks, one month, 2 months, and then as needed on a case-based basis. Outcomes of the treatment with oral antibiotics will be compared to the historical outcomes of patients treated with IV antibiotics at the University of Louisville oral and maxillofacial surgery clinic.

ELIGIBILITY:
The participant must meet each of the following inclusion criteria:

1. Clinical presentation of:

   1. localized pain OR
   2. localized erythema OR
   3. temperature >38.0ºC OR
   4. a discharging sinus or wound AND
2. willing and able to give informed consent AND
3. aged 18 years or above AND
4. the patient has received 7 days or less of intravenous therapy after an appropriate surgical intervention regardless of pre-surgical antibiotics
5. has a life expectancy > 1 year AND
6. has

   1. native osteomyelitis of the jaw (no hardware), either hematogenous or contiguous (odontogenic, trauma, etc) OR
   2. hardware or bone graft infection treated by debridement and retention, or by debridement and removal

   The exclusion criteria would consist of:
7. sepsis, septic shock, concomitant infection, or any need for prolonged hospitalization OR
8. tissue diagnosis other than "dead bone" OR
9. Staphylococcus aureus bacteremia on presentation or within a month OR
10. bacterial endocarditis on presentation or within the last 6 months OR
11. mild osteomyelitis not usually requiring prolonged IV antibiotics OR
12. when only IV form is available for a given antibiotic OR
13. the patient is unlikely to comply with trial OR
14. evidence of mycobacterial, fungal, parasitic, or viral etiology OR
15. participating in another clinical trial OR
16. pregnant patients OR
17. cognitively impaired patients or any situation in which informed consent cannot be obtained OR
18. incarcerated patients OR
19. patients with Chronic Nonbacterial Osteomyelitis (CNO) or Chronic Recurrent Multifocal Osteomyelitis (CRMO) OR
20. history of radiation to the jaws OR
21. history of bisphosphonate intake OR
22. patient less than 18 years of age

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-31 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Definite failure of antibiotic therapy in the treatment of orofacial osteomyelitis | 6-8 weeks
  The primary outcome will be a definite failure of antibiotic therapy indicated by one or more of the following (only resolution or failure will be recorded as the outcome):
  1. formation of a draining sinus tract arising from bone
  2. superficial spreading erythema, treated as cellulitis
  3. recurrence of frank pus
  4. no resolution of clinical signs and symptoms
  5. development of sepsis
  6. need for second surgery within 3 months (and if the first surgery is deemed adequate)
  7. recurrence of infection within 6 months

SECONDARY OUTCOMES:
Percentages of patients unable to complete treatment | 3-6 months
  Total number of patients that are unable to complete the proposed treatment due to any reason.
Patient Quality of life during therapy | 3-6 months
  Evaluate quality of life of patients receiving therapy. Quality of life will be evaluated by the EQ-5D assessment. Based on the results, the assessment is scored from 0-1. 1 represents the best possible health and 0 represents the worst possible health.
Treatment cost | 3-6 months
  Assessment of total monetary accumulation (in dollars $) per patient based on all interactions including the following: a) length of inpatient hospital stay, b) frequency of outpatient visits, c) inpatient and outpatient treatment costs
Incidence of Clostridium difficile associated diarrhea | 3-6 months
  Patients that develop the opportunistic infection clostridium difficile related to long term use of antibiotics for their treatment. Infection will be confirmed by stool sample.
Adherence | 3-6 months
  Adherence will be assessed by the Medication Event Monitoring Systems (MEMS) in participants. The MEMS system sensor in the pill bottle top detects opening and closing and records these events with a date stamp which helps verify whether patients accessed their bottles according to the schedule.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Louisville Oral and Maxillofacial Surgery Clinic, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes